CLINICAL TRIAL: NCT03811054
Title: The Efficacy and Drug Resistance Molecular Biology of Apatinib Combined With EGFR-TK1 Treated for Advanced Slow-progressed Non-Small Cell Lung Cancer (NSCLC)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Chest Hospital (Other)
Responsible Party: Principal Investigator, Liyan Xu, Chief of Medical Oncology Department, Beijing Chest Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BeijingCH002
Record Dates: First submitted 2019-01-14; First posted 2019-01-22 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Apatinib; Non Small Cell Lung Cancer; EGFR TKI; slowly progress
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Apatinib combined with EGFR-TKI (Experimental): Apatinib 250 millgram（mg/day（d））combined with EGFR-TKI
  Interventions: Drug: Apatinib（250mg/d） combined with EGFR-TKI

INTERVENTIONS:
Drug: Apatinib（250mg/d） combined with EGFR-TKI — Patients with advanced non-small cell lung cancer (NSCLC) who had treated with EGFR-TKI and progressed slowly because of resistance are underwent with apatinib mesylate and continuous EGFR-TKI.

SUMMARY:
Patients with advanced non-small cell lung cancer (NSCLC) who progress slowly after Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitors（EGFR-TKI）resistance. The purpose of this study is to investigate the efficacy and drug resistance mechanism of Apatinib combine with EGFR-TK1 treated for advanced slow progressed non-small cell lung cancer and provide new treatment options.

DETAILED DESCRIPTION:
Epidermal growth factor receptor Tyrosine kinase inhibitor (EGFR TKI) have been approved to treat NSCLC harboring EGFR mutation as first-line therapy. However, a large proportion of patients would become acquired resistant of EGFR-TKI after about one year although initially sensitivity. Previous studies demonstrated that the anti-angiogenesis combined with EGFR-TKI in slow-progressed EGFR mutation-positive non-small cell lung cancer achieved good efficacy and disease control rates, prolonged the progression free survival. The present study is aim to expand the number of samples to monitor resistance-related genes and tumor cells. Furthermore, to investigate the mechanism of anti-angiogenesis combine with EGFR-TKI and provide the theory for the use and promotion of clinically protocols. In this study, the primary objective is the objective response rates and the secondary goal are disease control rates, overall survival, progression free survival and drug safety.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent should be obtained before treatment. Patients with good compliance.
2. Histologically or cytologically confirmed IIIB/IV NSCLC.
3. Progress in the treatment of EGFR TKI.
4. Aged from 18 to 75 years (18 and 75 years are included); Gender Not Required.
5. ECOG PS 0-1.
6. Life expectancy ≥ 3 months.
7. At least one measurable lesion (meet the requirements of the standard Response Evaluation Criteria In Solid Tumors (RESCIST) version 1.1). If the lesions that have received local treatment (radiation, radiofrequency, intervention, etc.) are the only lesions, it is required to have clear imaging progress.

Exclusion Criteria:

1. Uncontrolled hypertension (systolic ≥140mmHg and/or diastolic ≥90mmHg after medication treatment); Poor control of blood sugar.
2. Acute phase of cerebral infarction, or recovery period <2 months.
3. A variety of factors that affect the absorption of oral medications (such as inability to swallow, nausea and vomiting, chronic diarrhea, intestinal obstruction, etc.)
4. Patients with a risk of gastrointestinal bleeding may not be enrolled, including the following: (1) active digestive ulcer lesions, and fecal occult blood (++); (2) a history of melena and hematemesis within 2 months. Simple fecal occult blood (+) is not an exclusion criterion.
5. Coagulation abnormality (INR>1.5×ULN, APTT>1.5×ULN), with bleeding tendency.
6. Urine protein ≥ ++ or confirmed 24-hour urine protein quantitation > 1.0 g.
7. Pregnant or lactating women.
8. Severe liver and kidney dysfunction (grade 4) .
9. Allergic to any ingredient of apatinib mesylate.
10. A history of abuse of psychotropic substances and are unable to quit smoking or mental disorders.
11. According to the investigator's judgment, people with concomitant diseases that seriously endanger the safety of the patient or affect the patient's completion of the study.
12. Surgery, major trauma or fracture, within 4 weeks before the treatment or unhealed wound before treatment.
13. Severe heart disease, such as grade III or above (NYHA standard) congestive heart failure, grade III or above (CCS standard) angina, a history of myocardial infarction within 6 months before the treatment, or medication treated arrhythmia.
14. Brain metastasis and meningeal metastasis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rates (ORR) | two years
  Objective response rate is defined as the percentage of subjects having achieved confirmed Complete Response + Partial Response according to Response Evaluation Criteria in Solid Tumors 1.1（RECIST1.1）

SECONDARY OUTCOMES:
Disease control rate (DCR) | two years
  Disease Control Rate is defined as the percentage of subjects having achieved confirmed Complete Response + Partial Response + Stable Disease according to radiological assessments.
Overall survival (OS) | two years
  Time from randomization to death for any cause.
Progression free survival (PFS) | two years
  PFS defined as date of randomization until the date of objectively determined progression defined by Response Evaluation Criteria in Solid Tumors criteria or death from any cause, whichever is first.
Drug safety: Number of participants with treatment-related adverse events | two years
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Locations (1):
- The Beijing Chest Hospital, Beijing, China